CLINICAL TRIAL: NCT06323902
Title: Clinical Evidence of Autologous Platelet-Rich Plasma as a Treatment for Macular Holes
Brief Title: Autologous Platelet-rich Plasma as a Treatment for Macular Holes
Status: Completed | Type: Observational
Sponsor: Clinica Oftalmologica Paredes (Other)
Responsible Party: Sponsor
Other Study IDs: PT-CO39
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Macular Holes; Macular Hole of Left Eye (Disorder); Macular Hole of Right Eye (Disorder)
Keywords: PLATELET RICH PLASMA; PLATELET GROWTH FACTORS; AUTOLOGOUS PLASMA; MACULAR HOLE
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with giant full thickness macular hole: 13 patients with a diagnosis of macular hole with a total thickness greater than 400 microns were chosen. Without prior vitreoretinal surgery
  Interventions: Procedure: Pars plana vitrectomy, with or without epiretinal membrane peeling, plus PRGF membrane implantation

INTERVENTIONS:
Procedure: Pars plana vitrectomy, with or without epiretinal membrane peeling, plus PRGF membrane implantation — In the operating room through pars plana vitrectomy after having completed the complete air exchange, with the help of a Backwash Charles cannula, the PRGF membrane is placed in the macular hole and C3F8 gas is left in the posterior chamber, the first hour in the recumbent position. supine and subsequently face down during the first postoperative week.
  Other Names: PRGF membrane implantation

SUMMARY:
For a series of patients with full-thickness macular hole, an autologous plasma rich in growth factors was developed in the form of a clot and applied to the retinal defect. These patients were followed up for a period of one year, obtaining substantial improvement both anatomically and functionally.

DETAILED DESCRIPTION:
A prospective observational study was carried out. Obtaining approval from the Institutional Ethics Committee at the Paredes Ophthalmology Clinic, in the city of Pasto - Colombia. This study adhered to the principles of the Declaration of Helsinki. 13 patients with a diagnosis of macular hole with a total thickness greater than 400 microns were chosen. The previous evaluation included a history and complete ophthalmological examination, uncorrected or better corrected visual acuity, optical coherence tomography - Optovue OCT and in some cases retinal photographs on the Eidon FA equipment. The inclusion criteria were: Patients without previous vitreoretinal surgery for macular hole, large full thickness macular hole.

During the consultation prior to scheduling the surgical procedure and on the day of the procedure, each patient was given a clear explanation about the intervention, doubts were resolved, and informed consent was signed in each case.

Following the institutional protocol for obtaining the platelet-rich plasma membrane, whole blood was obtained from each patient in 2 tubes with 3.2% sodium citrate, used as an anticoagulant. Subsequently, the samples were taken to be centrifuged at 3200 rpm for a period of 15 minutes, from here approximately 1.5 cc of plasma was obtained from each tube, without aspirating the white phase (leukocytes) or the red phase (erythrocytes), the plasma . obtained from each tube was placed in a single tube without anticoagulant and centrifuged again at 2700 rpm for a period of 7 minutes. Once the second centrifugation was completed, between 1 and 1.5 cc of the lower third of the plasma was obtained in a first syringe, to which 10% calcium gluconate was added with a ratio of 0.05 cc of calcium gluconate for every 1.5 cc plasma. Once the components are mixed, the plasma is spread with calcium gluconate on a petri dish forming a layer of approximately 2 mm. It is left covered at room temperature for approximately 30 minutes. The formation of clots in the layer is verified. plasma and went to the surgery room. The entire procedure was carried out under rigorous asepsis and sterility measures. In the operating room through pars plana vitrectomy after having completed the complete air exchange, with the help of a Backwash Charles cannula, the PRGF membrane is placed in the macular hole and C3F8 gas is left in the posterior chamber, the first hour in the recumbent position. supine and subsequently face down during the first postoperative week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of macular hole with a total thickness greater than 400 microns
* Patients without prior vitreoretinal surgery
* Patients over 18 years of age

Exclusion Criteria:

* Patients under 18 years of age
* Patients with previous vitreoretinal surgery
* Patients who had other additional retinal pathologies (diabetic retinopathy, hypertensive retinopathy, vascular retinal occlusions, retinal detachment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 13 patients were chosen with a diagnosis of macular hole with a total thickness greater than 400 microns, over 18 years of age, with no history of previous vitreretinal surgery or with other retinal pathologies. The triggering factors in 46% were due to the presence of an Epiretinal Membrane (6 cases) and 54% were due to vitreomacular traction (7 cases).
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Macular hole closure | Follow-up was carried out for 1 year
  The closure of the macular hole after PRGF membrane implantation was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Ofalmologica Paredes, Pasto, Departamento de Nariño, Colombia

IPD SHARING:
Plan to Share IPD: No
At the moment there is no plan to share the individual data of participants

REFERENCES:
- [Background] Majumdar S, Tripathy K. Macular Hole. 2023 Aug 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559200/ PMID 32644626
- [Background] Lyu WJ, Ji LB, Xiao Y, Fan YB, Cai XH. Treatment of refractory giant macular hole by vitrectomy with internal limiting membrane transplantation and autologous blood. Int J Ophthalmol. 2018 May 18;11(5):818-822. doi: 10.18240/ijo.2018.05.17. eCollection 2018. PMID 29862182
- [Background] Shen Y, Lin X, Zhang L, Wu M. Comparative efficacy evaluation of inverted internal limiting membrane flap technique and internal limiting membrane peeling in large macular holes: a systematic review and meta-analysis. BMC Ophthalmol. 2020 Jan 8;20(1):14. doi: 10.1186/s12886-019-1271-2. PMID 31914954
- [Background] Cisiecki S, Boninska K, Bednarski M. Autologous Lens Capsule Flap Transplantation for Persistent Macular Holes. J Ophthalmol. 2021 Feb 27;2021:8148792. doi: 10.1155/2021/8148792. eCollection 2021. PMID 33728059
- [Background] Buzzi M, Parisi G, Marolo P, Gelormini F, Ferrara M, Raimondi R, Allegrini D, Rossi T, Reibaldi M, Romano MR. The Short-Term Results of Autologous Platelet-Rich Plasma as an Adjuvant to Re-Intervention in the Treatment of Refractory Full-Thickness Macular Holes. J Clin Med. 2023 Mar 4;12(5):2050. doi: 10.3390/jcm12052050. PMID 36902837
- [Background] Okonkwo ON, Hassan AO, Akanbi T. Autologous Neurosensory Retinal Transplantation: A Report of Three Cases. J Ophthalmic Vis Res. 2021 Jan 20;16(1):68-76. doi: 10.18502/jovr.v16i1.8252. eCollection 2021 Jan-Mar. PMID 33520129
- [Background] Sanchez-Avila RM, Robayo-Esper CA, Villota-Deleu E, Fernandez-Vega Sanz A, Fernandez-Vega Gonzalez A, de la Sen-Corcuera B, Anitua E, Merayo-Lloves J. Plasma Rich in Growth Factors in Macular Hole Surgery. Clin Pract. 2022 Jan 10;12(1):57-69. doi: 10.3390/clinpract12010007. PMID 35076502
- [Background] Wang J, Rodriguez SH, Xiao J, Luo W, Gonnah R, Shaw L, Dao D, Schechet SA, Mackin AG, Komati R, Skondra D. FULL-THICKNESS MACULAR HOLE CLOSURE WITH TOPICAL MEDICAL THERAPY. Retina. 2024 Mar 1;44(3):392-399. doi: 10.1097/IAE.0000000000003988. PMID 37948745
- [Background] Galletero Pandelo L, Olaso Fernandez H, Sanchez Aparicio JA, Rodriguez Vidal C, Martinez-Alday N. Results of large macular hole surgery using different interposition techniques. A report on 9 cases. Arch Soc Esp Oftalmol (Engl Ed). 2022 Aug;97(8):457-463. doi: 10.1016/j.oftale.2022.03.010. Epub 2022 Mar 21. PMID 35331671
- See also: Macular Hole — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/32644626/
- See also: Treatment of refractory giant macular hole by vitrectomy with internal limiting membrane transplantation and autologous blood — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/29862182/
- See also: Comparative efficacy evaluation of inverted internal limiting membrane flap technique and internal limiting membrane peeling in large macular holes: a systematic review and meta-analysis — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/31914954/
- See also: Autologous Lens Capsule Flap Transplantation for Persistent Macular Holes — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/33728059/
- See also: The Short-Term Results of Autologous Platelet-Rich Plasma as an Adjuvant to Re-Intervention in the Treatment of Refractory Full-Thickness Macular Holes — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/36902837/
- See also: Autologous Neurosensory Retinal Transplantation: A Report of Three Cases — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/33520129/
- See also: Plasma Rich in Growth Factors in Macular Hole Surgery — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/35076502/
- See also: FULL-THICKNESS MACULAR HOLE CLOSURE WITH TOPICAL MEDICAL THERAPY — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/37948745/
- See also: Results of large macular hole surgery using different interposition techniques. A report on 9 cases — https://pubmed-ncbi-nlm-nih-gov.udea.lookproxy.com/35331671/